CLINICAL TRIAL: NCT02511717
Title: A Randomized Trial of Transcutaneous Nerve Stimulation for Overactive Bladder Patients
Brief Title: A Trial of Transcutaneous Nerve Stimulation for OAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Blayne Welk, Assistant Professor of Surgery, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 106903
Record Dates: First submitted 2015-07-28; First posted 2015-07-30 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham (Sham Comparator): Transcutaneous stimulation in a location and with settings not relation to the bladder nerves, 3x/week for 30 minutes for 12 weeks
  Interventions: Other: Sham transcutaneous tibial nerve stimulation
- Transcutaneous nerve stimulation (Active Comparator): Transcutaneous stimulation of the bladder nerves, 3x/week for 30 minutes for 12 weeks
  Interventions: Other: Transcutaneous tibial nerve stimulation

INTERVENTIONS:
Other: Transcutaneous tibial nerve stimulation — Patch electrodes applied posterior to the medial malleolus, and 5-10 cm above the medial malleolus of the same leg, just behind the medial tibial edge. Bipolar stimulation setting will be used, with a frequency of 10 Hz, 200ms pulse, and the amplitude will be titrated up to patient's maximum nonpainful tolerance (between 0.5-10mA). This will be done by the patients at home 3x/week for 30 minutes, over 12 weeks.
  Arms: Transcutaneous nerve stimulation
Other: Sham transcutaneous tibial nerve stimulation — Patch electrodes applied posterior to the lateral malleolus, and 5-10 cm above the lateral malleolus of the same leg. Bipolar stimulation setting will be used, with a frequency of 10 Hz, 200ms pulse, and the amplitude will be set a 1mA. This will be done by the patients at home 3x/week for 30 minutes, over 12 weeks.
  Arms: Sham

SUMMARY:
Overactive bladder causes urinary frequency, urgency and in some cases urgency incontinence. This study is testing the efficacy of transcutaneous tibial nerve stimulation (using skin patch electrodes via a transcutaneous electrical nerve stimulation (TENS) machine) for the treatment of women with clinical symptoms of overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

1. Female, >18 years of age, with the clinical diagnosis of overactive bladder.
2. Failure of behavioral measures and pharmacologic therapy to adequately control overactive bladder symptoms.
3. Baseline patient perception of bladder condition score of 2 or higher.

Exclusion Criteria:

1. Current or previous percutaneous or sacral neuromodulation therapy
2. Stress predominant urinary incontinence
3. Newly added bladder medication or dose change with the last 2 months (Tamsulosin, Silodosin, Alfuzosin, Terazosin, Baclofen, Diazepam, amitriptyline, imipramine, DDAVP, tolterodine, oxybutynin, fesoterodine, darifenacin, solifenacin, trospium, mirabegron)
4. Intravesical botulinum toxin use within the last 1 year
5. Implanted pacemaker or defibrillator
6. History of epilepsy
7. Unable or unwilling to commit to study treatment schedule
8. Pregnant, or possible pregnancy planned for the duration of the study period
9. Active skin disease of the lower legs (dermatitis, cellulitis, eczema, trauma)
10. Documented allergy to patch electrodes or their adhesive
11. Abnormal sensory function of the lower limb
12. Metallic implant within the lower limb

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St Josephs Health Care, London, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham | Transcutaneous Nerve Stimulation
Started | 10 | 10
Completed | 8 | 10
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham | Transcutaneous Nerve Stimulation | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [58 to 67] | 64 [59 to 70] | 64 [59 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Outcome Measure (Patient Percention of Bladder Condition Question)
Description: Patient percention of bladder condition (PPBC) question. It is scored from 0 (My bladder condition does not cause me any problems at all) to 5 (My bladder condition causes me many severe problems). Higher numbers are worse outcomes.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Sham | Transcutaneous Nerve Stimulation
Number analyzed (Participants) | 10 | 10
units on a scale | 4 [3 to 5] | 3 [2 to 4]

2. Secondary Outcome: Overactive Bladder Questionnaire Short Form (OAB-q SF)
Description: OAB quality of life questionnaire
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Voiding Diary
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: 24hr Pad Weights
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Physician Assessment of Treatment Benefit
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Sham | Transcutaneous Nerve Stimulation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT02511717/Prot_SAP_000.pdf